CLINICAL TRIAL: NCT04053712
Title: Dual-hormone Closed-loop Glucose Control in Type 1 Diabetes
Acronym: DHCL2019
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Steno Diabetes Center Copenhagen (Other)
Collaborators: Technical University of Denmark (Other); University of Copenhagen (Other); Danish Diabetes Academy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: H-19026331; 2019-001631-31 (EudraCT Number); 2019043528 (Registry Identifier: Danish Medical Agency); 2019043269 (Registry Identifier: Danish Medical Agency - Device regulation); CIV-19-04-028465 (Registry Identifier: CIV ID)
Record Dates: First submitted 2019-08-08; First posted 2019-08-12 (Actual); Last update posted 2022-08-18 (Actual); Status verified 2022-08

CONDITIONS: Type 1 Diabetes; Hypoglycemia
Keywords: Closed-loop; Dual-hormone; Glucagon; FiAsp; Artificial pancreas
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Hypoglycemia | interventions — Glucagon

STUDY DESIGN:
Intervention Model Description: A randomized single-blinded placebo-controlled cross-over 33-hour in-clinic study in adults with type 1 diabetes.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Single-hormone (Placebo Comparator): FiAsp (R) - Saline
  Interventions: Device: Closed-loop system
- Dual-hormone (Active Comparator): FiAsp(R) - GlucaGen(R)
  Interventions: Drug: Glucagon; Device: Closed-loop system

INTERVENTIONS:
Drug: Glucagon — GlucaGen(R), Novo Nordisk, DK
  Arms: Dual-hormone
Device: Closed-loop system — Closed-loop system comprise of two DANA RS (R) insulin pumps (FiAsp-GlucaGen vs FiAsp-saline), one DexCom G6 sensor, and a smartphone for the control algorithm.

SUMMARY:
Despite recent pharmacological and technological advantages, hypoglycemia remains to be the key limiting factor in achieving optimal glycemic control in people with type 1 diabetes. State-of-the-art treatment for type 1 diabetes is insulin in pens or pumps that focus on reducing hyperglycemia after relative insulin deficiency e.g. after food intake. In recent years, we focused on adding low-dose glucagon to insulin therapies for the treatment and prevention of hypoglycemia - referred to as "dual-hormone treatment". We have shown that low-dose glucagon is efficient in treating mild hypoglycemia and that several factors may affect its glucose response. Our next step is to test whether the combined delivery of insulin and glucagon can improve glucose control in individuals with type 1 diabetes. In this proposal, we want to test the efficacy, safety and feasibility of a dual-hormone closed-loop system, also known as an artificial pancreas. The closed-loop system involves automatic infusion of glucagon and insulin based on continuous glucose measurements. The system will be tested in a 33-hour in-clinic study comparing the glucose control by the combined automatic delivery of insulin and glucagon with the automatic delivery of insulin-only. The study is performed at Steno Diabetes Center Copenhagen (SDCC) in collaboration with the Technical University of Denmark (DTU). We expect that the study will clarify whether low-dose glucagon added to insulin therapy can improve the glucose control in adults with type 1 diabetes. We believe that the utilization of glucagon will allow for a weight neutral optimization of glucose control, reduce risk of hypoglycemia and reduce disease burden that will reduce diabetes complications and cardiovascular diseases.

DETAILED DESCRIPTION:
Rationale: We hypothesize that our newly developed dual-hormone insulin-glucagon closed-loop system (DCL) is safe, efficient and superior to our single-hormone insulin-only closed-loop system (SCL). The study aims to compare the glucose control achieved by DCL with our SCL.

Design: A randomized single-blinded placebo-controlled cross-over 33-hour in-clinic study of glucose control achieved with DCL versus SCL in adults and adolescents with type 1 diabetes.

Participants: 13 insulin-pump treated T1D participants will be included, if they are 15-80 years old, have T1D for ≥ 3 years, use insulin pumps with FiAsp®, and have an HbA1c≤ 8.5% (69 mmol/mol).

Procedures: In this two-phase study 1) we test the operability of our closed-loop systems and 2) compare glucose control by DCL with SCL. The two studies are identical except for the blinding procedures. In the first phase (pilot study), four participants are included, and the glucagon/saline pump is not masked. In the second phase (main study), 13 participants are included, and are as well as the investigators blinded for the content in the glucagon/saline pump.

Two days prior to study visit, a CGM (Dexcom® G6) is place on the participant's abdomen. At study visits, participants arrive in the evening at our research unit and get their insulin pump disconnected. Two study pumps (Dana Diabecare RS®, SOOIL) are attached: one pump infuses insulin (FiAsp®, Novo Nordisk) and the other infuses either glucagon (GlucaGen®, Novo Nordisk) or saline. Once a sampling cannula is placed in an antecubital vein, the study is initiated and the closed-loop system (DCL vs SCL) takes over the glucose control for the next 33 hours. Except from the control algorithm (SCL vs DCL), the study days are identical. Participants can move around freely in the clinic for 33 hours but will perform a 45-min moderate (50% VO2max) exercise session, consume three meals with variant carbohydrate content, and sleep during two overnight periods. Participants will be monitored frequently with blood samples (drawn from the antecubital vein), blood pressure, pulse, and VAS scale for nausea.

ELIGIBILITY:
Inclusion criteria

* Age ≥ 18 years
* T1D ≥ 2 years
* Insulin pump therapy ≥ 1
* Currently treated with FiAsp® - insulin
* HbA1c ≤ 8.5% (69 mmol/mol) Exclusion criteria
* Pregnancy or nursing
* Inability and willingness to comply with all protocol procedures, e.g. exercise, sleeping, blood sampling, and meal consumption
* Plan to become pregnant or sexually active and not using adequate contraceptive methods (sterilization, intrauterine device, contraceptive pill, patch or injection)
* Hypoglycemia unawareness (self-reported lack of hypoglycemia symptoms when blood glucose is < 3.0 mmol/l)
* Use of anti-diabetic medicine (other than insulin), corticosteroids or other drugs affecting glucose metabolism during or within 30 days prior to study participation
* History of coronary artery disease or congestive heart failure
* Abnormal ECG suggestive of coronary artery disease and increased risk of malignant arrhythmia
* Allergy to glucagon or lactose
* Pheochromocytoma
* Other concomitant medical or psychological condition that according to the investigator's assessment makes the patient unsuitable for study participation

Withdrawal criteria

* In case of pregnancy (or desire for pregnancy), female subjects are withdrawn
* Lack of compliance to any of the important study procedures in the discretion of the investigator
* Unacceptable adverse effects in the discretion of the investigator
* Withdrawal on participants request will be accepted at any time without further justification

Patients who complete or withdraw from the study continue their usual quarterly follow-up visits at the diabetes clinic. Withdrawal does not affect their statutory patient rights.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 13 (Actual)
Dates: Start 2019-07-16 (Actual); Primary Completion 2021-03-19 (Actual); Study Completion 2021-03-19 (Actual)

PRIMARY OUTCOMES:
Percentage of time with glucose values < 3.9 mmol/l as measured by glucose sensor | 33 hours
Number of carbohydrate interventions to treat hypoglycemia | 33 hours
  Carbohydrate interventions are predefined and provided in case of hypoglycemia

SECONDARY OUTCOMES:
Percentage of time with glucose values < 3.9 mmol/l as measured by venous plasma glucose | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Percentage of participants achieving (A) time in range (3.9-10 mmol/l) > 70 %, (B) time in alert hypoglycemia (<3.9 mmol/l) < 4 %, and (C) time in clinical hypoglycemia (<3.0 mmol) < 1% as measured by glucose sensor and venous plasma glucose | 33 hours
  A composite outcome will be calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Mean blood glucose value measured by glucose sensor and venous plasma glucose | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Percentage of time with glucose values in the range 3.9-8.0 mmol/l measured by glucose sensor and venous plasma glucose | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Percentage of time with glucose values in the range 3.9-10.0 mmol/l measured by glucose sensor and venous plasma glucose | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Percentage of time with glucose values in the range > 13.9 measured by glucose sensor and venous plasma glucose | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Percentage of time with glucose values < 3.0 mmol/l as measured by glucose sensor and venous plasma glucose | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Number of hypoglycemic episodes (<3.9 mmol/l and <3.0 mmol/l) overnight and during daytime | 33 hours
Nadir blood glucose value for each hypoglycemic episode as measured by glucose sensor and venous plasma glucose | 33 hours
Glucose sensor glycemic variability measured as SD and CV during overnight and during daytime | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Low Blood Glucose Index (LBGI) overnight and during daytime by glucose sensor and venous plasma glucose | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Percentage of participants with a mean blood glucose value (glucose sensor and venous plasma glucose) ≤ 8.6 mmol/l (corresponding to an estimated HbA1c of 7.0% / 53 mmol/mol) | 33 hours
Percentage of patients with a mean blood glucose value (glucose sensor and venous plasma glucose) ≤ their standard therapy mean glucose value (calculated based on HbA1c measurement) | 33 hours
Mean Absolute Relative Difference (MARD) between glucose sensor and venous plasma glucose | 33 hours
  Participants have two glucose sensors during the study
Percentages of values between glucose sensor and venous plasma glucose in zone A, B, C, D and E in the Clarke Error Grid analysis. | 33 hours
  Participants have two glucose sensors during the study. One sensor closed to the infusion of glucagon.
Mean blood pressure over the study period (mmHG) | 33 hours
  Blood pressure and pulse taken at predefined timepoints
Mean pulse rate over the study period (beats per min) | 33 hours
  Blood pressure and pulse taken at predefined timepoints
Mean nausea level measured with a visual analog scale (VAS range: 0-10) | 33 hours
  Calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Total insulin dose per study day (UI) | 33 hours
Total time of insulin suspension per study day (UI) | 33 hours
Total glucagon dose per study day (microgram) | 33 hours
  the outcome will be calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Mean plasma glucagon | 33 hours
  the outcome will be calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Mean plasma insulin aspart | 33 hours
  the outcome will be calculated for the whole study period as well as for the following intervals: night 1 (23:00-07:00), night 2 (23:00-07:00), night 1 and 2, 23:00-15:00 and 15:00-07:00.
Difference in participant estimated grams of carbohydrate and actual carbohydrate in study meals | 33 hours
  Meals presented at the study will be estimated for carbohydrate content by the participant on
Difference in participant estimated blood glucose level and plasma glucose level at predefined timepoints | 33 hours
  Self-assessment of glucose levels (Clarke Error Grid)
Total energy expenditure during the study visit (kcal/kg) measured by ActiGraph GT9X Link | 33 hours
  Freedson and Sasaki MET prediction equations to determine energy expenditure in MET
Steps taken during the study visit measured by ActiGraph GT9X Link | 33 hours
Minutes per study day (min/d) spent in different levels of activity (sedentary, light, moderate, vigorous, or MVPA) measured by ActiGraph GT9X Link | 45 min
Minutes between lights off and the first sleep episode (Sleep latency) measured by ActiGraph GT9X Link | 14 hours
Total sleep time measured by ActiGraph GT9X Link | 14 hours
  Minutes between sleep onset and wake time
The percentage of time asleep from lights off to lights on (sleep efficiency) measured by ActiGraph GT9X Link | 14 hours
Mean Borg scale level during exercise (RANGE:0-10) | 45 min
  Assessed every 5-10 minutes during bicycling

CONTACTS AND LOCATIONS:
Overall Officials: Ajenthen G Ranjan, MD, PhD, Principal Investigator — Steno Diabetes Center Copenhagen
Locations (1):
- Steno Diabetes Center Copenhagen, Gentofte Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, CSR